CLINICAL TRIAL: NCT03670823
Title: A Combination of Innovative Technologies: EEG, Eye Tracking Device and fMRI in Order to Predict the Success of SSRI Treatment in Patients With Major Depression.
Brief Title: Prediction of SSRI Treatment in Major Depression.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ElMindA Ltd (Industry)
Collaborators: Sheba Medical Center (Other Government); Hebrew University of Jerusalem (Other)
Responsible Party: Sponsor
Other Study IDs: ELM-55 5323-18-SMC
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-05

CONDITIONS: Major Depression
Keywords: Major Depression; EEG; Eye Tracker; fMRI; MRI; Resting State Connectivity; Cognition
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Healthy subjects: 50 healthy subjects for a control group
  Interventions: Device: SIEMENS PRISMA MRI
- Patients with Major Depression: 50 patients with major depression for a research group
  Interventions: Device: SIEMENS PRISMA MRI

INTERVENTIONS:
Device: SIEMENS PRISMA MRI — Collect data on brain activation from different methods
  Other Names: BNA (EEG) Technology, Eyetracking device

SUMMARY:
This project will combine the data collected from EEG, Eye tracking, structural and functional MRI scans and neuropsychological performance from patients with major depression receiving SSRI treatment. The purpose of this research is to predict the success of the SSRI treatment and to categorize patients into sub-groups according to similar patterns of brain activation to personalize treatment.

DETAILED DESCRIPTION:
Major depression is a mood disorder affecting 350 million people worldwide. The disorder is characterized by depressed mood, anhedonia, decreased quality of life, deficits in cognitive functions and even suicide thoughts. Treatment of depression is often a long process and includes taking different types and quantities of medications. Therefore, there is a need to predict the success of the SSRI treatment. Our research will examine the outcomes of the combined technologies: BNA (EEG), Eye-tracker, structural and functional MRI scans and neuropsychology tasks in patients with depression while receiving SSRI treatment. The purpose of the research is to track biomarkers and other measures, which will allow predicting the SSRI treatment's success within 4 weeks instead of 8 weeks. In addition, the investigators will attempt to categorize patients into different subgroups according to their brain activation and eye movements. This division into subgroups may contribute to the understanding of the mechanisms that account for the responsiveness to SSRI treatment and to the possibility of targeting patients with depression towards a particular treatment. From this research, the investigators aim to personalize the treatment of depression, make it more efficient and reduce the amount of time for the patient to reach an optimal responsiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-65 years old
2. Male and female
3. Ability to comprehend and sign informed consent
4. DSM-5 diagnosis with MINI 7.0.2 (healthy subjects need to be ruled out)

Inclusion Criteria for patients with depression:

1. DSM-5 diagnosis
2. 0-2 failed treatments
3. Patients which will start SSRI treatment

Exclusion Criteria:

1. unconsciousness
2. Pregnancy or nursing
3. Cardiovascular instability
4. Metabolic instability (water, electrolytes, sugar)
5. Fever or evidence of microbiological pollutant
6. Deafness or blindness
7. Schizophrenia
8. Addiction disorders
9. Eating disorders
10. Bi-polar disorder
11. Cognitive deficits
12. Start a new psychotherapy during the research
13. Unable to enter the MRI scanner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will include 2 groups of subjects: healthy subjects and patients with major depression
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
EEG responses to cognitive tasks in combination with the Eye-tracker Device. | 2 years
  Categorize patients into subgroups according to combined measures of EEG and Eye

SECONDARY OUTCOMES:
Resting state connectivity analysis | 2 years
  Examine the difference in resting state connectivity between the groups.
Examine correlations between the different methods | 2 years
  Examine correlations between the different methods EEG, Eye-tracking and fMRI
EEG brain activation to cognitive tasks | 2 years
  Categorize patients into subgroups according to similar brain activity
Eye-tracking tasks | 2 years
  Categorize patients into subgroups according to similar patterns of eye movements.
Examine MRI structural changes | 2 years
  Compare structural changes between the groups (patients with depression, healthy subjects).
Cognitive scores on CANTAB (computerized cognitive assessments) | 2 years
  Examine the difference in responses to different cognitive exams between the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical CENTER, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drysdale AT, Grosenick L, Downar J, Dunlop K, Mansouri F, Meng Y, Fetcho RN, Zebley B, Oathes DJ, Etkin A, Schatzberg AF, Sudheimer K, Keller J, Mayberg HS, Gunning FM, Alexopoulos GS, Fox MD, Pascual-Leone A, Voss HU, Casey BJ, Dubin MJ, Liston C. Resting-state connectivity biomarkers define neurophysiological subtypes of depression. Nat Med. 2017 Jan;23(1):28-38. doi: 10.1038/nm.4246. Epub 2016 Dec 5. PMID 27918562
- [Background] Ogawa T, Sekino H, Uzura M, Sakamoto T, Taguchi Y, Yamaguchi Y, Hayashi T, Yamanaka I, Oohama N, Imaki S. Comparative study of magnetic resonance and CT scan imaging in cases of severe head injury. Acta Neurochir Suppl (Wien). 1992;55:8-10. doi: 10.1007/978-3-7091-9233-7_3. PMID 1414552
- [Background] Raichle ME, Snyder AZ. A default mode of brain function: a brief history of an evolving idea. Neuroimage. 2007 Oct 1;37(4):1083-90; discussion 1097-9. doi: 10.1016/j.neuroimage.2007.02.041. Epub 2007 Mar 6. PMID 17719799
- [Background] Rohden AI, Benchaya MC, Camargo RS, Moreira TC, Barros HMT, Ferigolo M. Dropout Prevalence and Associated Factors in Randomized Clinical Trials of Adolescents Treated for Depression: Systematic Review and Meta-analysis. Clin Ther. 2017 May;39(5):971-992.e4. doi: 10.1016/j.clinthera.2017.03.017. Epub 2017 May 2. PMID 28476404